CLINICAL TRIAL: NCT03026621
Title: Examining the Change in Microbiome Diversity and Urine Metabolites After Lignite Extract Use
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seraphic Group Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 104
Record Dates: First submitted 2017-01-17; First posted 2017-01-20 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Microbiome
MeSH Terms: interventions — Coal; Teas, Herbal

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator): This will be an herbal tea the looks similar to the control.
  Interventions: Other: Herbal tea
- Lignite Extract (Experimental): This will be the Restore gut supplement
  Interventions: Dietary Supplement: Lignite Extract

INTERVENTIONS:
Dietary Supplement: Lignite Extract — The study design is a double-blind case-control trial, whereby half of the participants will be "cases" and will be asked to take 5mL 'Restore' mineral supplement three times each day. The other half of the participants will be "controls" and will be asked to take 5mL of a placebo three times each day. Both the study leader and the participants will be blinded to who receives Restore and who receive placebo.
  Other Names: Restore Gut Supplement
  Arms: Lignite Extract
Other: Herbal tea — This is an herbal tea that will look like the control
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether or not 'Restore' lignite extract mineral supplement impacts the microbiome composition of the mouth and gut. Additionally, participant urine samples will be examined to determine whether or not 'Restore' mineral supplement impacts the composition urine biomarkers and toxins.

DETAILED DESCRIPTION:
OBJECTIVES:

The purpose of this study is to determine whether or not 'Restore' lignite extract mineral supplement impacts the microbiome composition of the mouth and gut. Additionally, participant urine samples will be examined to determine whether or not 'Restore' mineral supplement impacts the composition urine biomarkers and toxins.

BACKGROUND & RATIONALE There is mounting evidence that the composition of the microbiome can change quickly. Unpublished case reports have shown significant shifts in the microbiome when participant's diet changes from a high carbohydrate to a high fat diet. Clinically, the use of 'Restore' mineral supplement has led to the bulking of stool in people using it for the first time within one or two days of first dose, further indicating a change in the gut microbiome.

Given these observations, this clinical trial was designed to examine how taking 'Restore' mineral supplement may impact the microbiome by examining the gut bacteria composition at two days, and again at two weeks. Our hypothesis is that taking Restore alone can lead to a quantifiable shift in the diversity of the microbiome as measured by the Simpson's Diversity Index, a mathematical measure of species diversity in a community. This index provides more information about community composition than simply species richness by also taking into account the relative abundances of different species.

There is also evidence that Restore mineral supplement can impact urine composition. Specifically, we will be examining the change in the presence of zonulin, glyphosate, creatinine-albumin ratio, and stem cells.

ELIGIBILITY:
Inclusion Criteria:

* People over 18 and under 80 who have never taken Restore gut supplement

Exclusion Criteria:,

* pregnant women, prisoners, people with primary bowel disorder or who have taken antibiotics over the last four weeks

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Intestinal Microbiome | 2 weeks
  Next generation genetic sequence will be taken

SECONDARY OUTCOMES:
Oral Microbiome | 2 weeks
  Next generation genetic sequence will be taken
Urine metabolies | 2 weeks
  Urine glyphosate, CD34, zonulin, creatine-albumin ratio and a urine analysis panel

CONTACTS AND LOCATIONS:
Overall Officials: David Roberts, Principal Investigator — Seraphic Group
Locations (1):
- Biomic Sciences, Charlottesville, Virginia, United States